CLINICAL TRIAL: NCT05691959
Title: Calcium Administration to Prevent Hypotension Caused by Diltiazem Administration in the Treatment of Atrial Fibrillation With Rapid Ventricular Response
Brief Title: Pre-diltiazem, Calcium Versus Placebo for Atrial Fibrillation With Rapid Ventricular Response
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ascension Health (Industry)
Responsible Party: Principal Investigator, Virginia LaBond MD, Core Faculty/Research Advisor, Emergency Medicine Residency Program, Ascension Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RMI20220086
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation With Rapid Ventricular Response; Hypotension
Keywords: Atrial Fibrillation; Rapid Ventricular Response; Diltiazem; Calcium Channel Blocker; Calcium; Hypotension; Heart Rate
MeSH Terms: conditions — Hypotension; Atrial Fibrillation | interventions — Saline Solution; Calcium; Drug Evaluation

STUDY DESIGN:
Intervention Model Description: Randomized Placebo Controlled Double Blind Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each formulation is masked by the pharmacy department.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Normal Saline (Placebo Comparator): Normal saline 50 ml intravenous piggyback once over 10 minutes
  Interventions: Drug: Placebo
- Calcium chloride (Experimental): x grams in 50 ml ivpb once over 10 minutes
  Interventions: Drug: Calcium

INTERVENTIONS:
Drug: Placebo — Patients randomized to placebo group will receive Normal Saline 50ml IV.
  Other Names: Normal saline
  Arms: Normal Saline
Drug: Calcium — Patients randomized to the study group will receive Calcium 2gm in Normal Saline 50ml IV.
  Other Names: Study drug
  Arms: Calcium chloride

SUMMARY:
The goal of this randomized double blind controlled trial is to learn about the effects of calcium when it is given prior to diltiazem for patients with atrial fibrillation ( a type of irregular heart beat) who have rapid ventricular response ( a pulse over 100 beats per minute). Normally diltiazem 0.25mg/kg (max 20mg) is given to slow the heart rate. We will give Placebo versus Calcium Gluconate 2gm given prior to diltiazem.

The main questions it aims to answer are:

* Does calcium decrease the incidence of low blood pressure (a side effect of diltiazem)?
* How does calcium effect the action of diltiazem? Does it interfere with the desired decrease in heart rate?

Participants will receive either placebo or calcium immediately prior to the administration of diltiazem. Their blood pressure and pulse will be measured:

* prior to study drug administration
* post study drug and prior to diltiazem administration
* 3 minutes post start of diltiazem
* 5 minutes post start of diltiazem
* 10 minutes post start of diltiazem
* 20 minutes post start of diltiazem
* 30 minutes post start of diltiazem

Researchers will compare the placebo group to the calcium group to see if there is a difference in the blood pressure and pulse.

DETAILED DESCRIPTION:
Diltiazem, a calcium channel blocker is the standard of care for treatment of stable patients with atrial fibrillation and rapid ventricular response. Many emergency physicians opine that calcium, the "antidote" for calcium channel blockers, when given prior to diltiazem administration, mitigates the common adverse effect of hypotension.

In order to obtain evidence related to this belief, we will study the effects of placebo (normal saline 50ml) versus calcium gluconate (2 grams in normal saline 50ml). Hemodynamically stable patients in afib with rvr will be identified on their arrival to the emergency department. Those who consent to the study will be enrolled and the pharmacy will be contacted to provide a blinded study sample to the patient's bedside. After initial vital signs are recorded the study sample will be infused via pump over a 10 minute period. Vitals will be recorded on its completion and a diltiazem bolus (0.25mg/kg, max 20mg) will be administered. Vitals will be recorded at 3, 5, 10, 20 and 30 minutes post start of diltiazem bolus.

The primary outcome of hypotension will be calculated using rates (frequencies). The rate of hypotension will be compared between the two groups using Chi square analysis. The groups will be compared for similarity using means(sd) and frequencies(percentages). Any variables that differ by group will be controlled for with a multiple logistic regression analysis.

A 35% rate of hypotension is estimated for the placebo group and a hypothesized 22% in the treatment group (a relative 37% decrease). This will require a minimum total sample size of 378 (184/ group) . We may terminate the study earlier if we achieve power.

ELIGIBILITY:
Inclusion Criteria: Diagnosis of atrial fibrillation with rapid ventricular response (ventricular rate over 100 bpm) due to an electrophysiologic etiology.

-

Exclusion Criteria:

1. Unstable, requiring electric cardioversion -hypotensive

   * altered mental status
   * myocardial infarction
   * pulmonary hypertension
2. Patients at risk of hypercalcemia - renal failure
3. Know cardiac valvular disease
4. Allergic to calcium gluconate or diltiazem
5. Underlying cardiac disease - sick sinus syndrome

   * 2nd/3rd degree atrial ventricular block
   * cardiogenic shock
   * recent IV beta blocker administration
   * accession bypass tract (WPW, short PR)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2023-01-26 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Hypotension | Thirty minutes from time of drug administration
  Mean arterial blood pressure less than 70mm Hg

SECONDARY OUTCOMES:
Heart rate | Thirty minutes from drug administration
  Decrease below 100 beats per minute

CONTACTS AND LOCATIONS:
Overall Officials: Virginia A LaBond, MS MD, Principal Investigator — Ascension Health

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Barnett JC, Touchon RC. Short-term control of supraventricular tachycardia with verapamil infusion and calcium pretreatment. Chest. 1990 May;97(5):1106-9. doi: 10.1378/chest.97.5.1106. PMID 2331904
- [Background] Haft JI, Habbab MA. Treatment of atrial arrhythmias. Effectiveness of verapamil when preceded by calcium infusion. Arch Intern Med. 1986 Jun;146(6):1085-9. doi: 10.1001/archinte.146.6.1085. PMID 3718093
- [Background] Kolkebeck T, Abbrescia K, Pfaff J, Glynn T, Ward JA. Calcium chloride before i.v. diltiazem in the management of atrial fibrillation. J Emerg Med. 2004 May;26(4):395-400. doi: 10.1016/j.jemermed.2003.12.020. PMID 15093843
- [Background] Lee J, Kim K, Lee CC, Nam YW, Lee JH, Rhee JE, Singer AJ, Kim KS, Ro Y. Low-dose diltiazem in atrial fibrillation with rapid ventricular response. Am J Emerg Med. 2011 Oct;29(8):849-54. doi: 10.1016/j.ajem.2010.03.021. Epub 2010 May 1. PMID 20825912
- [Background] Moser LR, Smythe MA, Tisdale JE. The use of calcium salts in the prevention and management of verapamil-induced hypotension. Ann Pharmacother. 2000 May;34(5):622-9. doi: 10.1345/aph.18318. PMID 10852091
- See also: rate control therapy — https://www.uptodate.com/contents/control-of-ventricular-rate-in-atrial-fibrillation-pharmacologic-therapy?sear
- See also: calcium gluconate drug information — http://www.uptodate.com/contents/calcium-gluconate-drug-information?search=calcium+gluconate&source=pa
- See also: diltiazem drug information — http://www.uptodate.com/contents/diltiazem-drug-information?source=history_widget